CLINICAL TRIAL: NCT01750658
Title: ECOS: A Study of Chronic Obstructive Pulmonary Disease (COPD) Exacerbations In Spain (o Estudio de Las Exacerbaciones de la EPOC en España)
Brief Title: Study of Chronic Obstructive Pulmonary Disease (COPD) Exacerbations In Spain
Acronym: ECOS
Status: Completed | Type: Observational
Sponsor: Cimera (Network)
Collaborators: Hospital Son Espases (Other); HOSPITAL DOCE DE OCTUBRE (Unknown); Hospital Clinic of Barcelona (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital La Fe de Valencia (Unknown); Hospital de Galdakao (Other); Hospital del Mar (Other)
Responsible Party: Sponsor
Other Study IDs: Nº IB 497/05
Record Dates: First submitted 2012-11-14; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: COPD
Keywords: Biomarkers; Exacerbations; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: COPD patients admitted in any of the participating ECOS hospitals due to a COPD exacerbation.
  1. - External factors. The episodes of COPD exacerbations are associated to exogenous factors (pollution, change of ambient temperature, humidity, infections). The prevalence of environmental contamination and infections is higher than expected.
  2. - Endogenous factors. These factors (hyperinflation, pulmonary embolism, cardiac dysfunction, mucus hypersecretion) are present in a proportion higher than expected
  3. - During exacerbations of COPD serum markers of inflammation and autoimmunity are high relative to baseline in COPD and decrease progressively during the follow-up, after controlling the acute episode

SUMMARY:
ECOS is a cross-sectional, observational, longitudinal, multicenter study enrolling 100-200 patients during a COPD exacerbation.

DETAILED DESCRIPTION:
Patients will be followed for 12 months. Information to be collected includes clinical, analytical, immunological, microbiological, hemodynamic, imaging, environmental, social and other blood markers of inflammation (IL-8, IL-6, TNF, TNF-alpha, endothelin-1, SLPI, IL10, TGF-beta and markers oxidative stress (TEAC)), and sputum (cell count, IL-6, IL-8, SLPI, ET 1, IL10).

Each center will collect clinical data, blood gas, microbiological and functional data for their patients, which will be centralized through the website of the Red Respira (www.redrespira.net).

A frozen serum sample and another of frozen sputum supernatant will be sent to the coordinating center (Palma de Mallorca).

Statistical analysis will include descriptive statistics: mean, standard deviation and range. Comparison of quantitative variables to be assessed using Student's t-test and ANOVA. Correlations between variables will be performed using bivariate analyzes (Pearson's linear correlation coefficient) and multivariate (multiple regression) analyses, among others.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 40-80 years
* Diagnosis of COPD (according to ATS/ERS consensus guidelines)
* Smoking history ≥ 10 pack years
* Hospitalization for exacerbation of COPD

Exclusion Criteria:

* Pneumonia.
* Pneumothorax.
* Severe comorbidities, such as:
* -Advanced cancer.
* -Pulmonary tuberculosis, which affects more than one third of the total lung parenchyma.
* -Pneumonectomy.
* -Previous diagnosis of left heart failure.
* -Cardiomyopathy with ventricular dysfunction (ejection fraction <45%).
* -Chronic inflammatory diseases such as asthma, rheumatoid arthritis, pulmonary fibrosis and autoimmune diseases.
* Mechanical Ventilation.
* Existence of an exacerbation of COPD in the 4 weeks prior to admission.
* MRSA.
* History of thoracic/lung surgery in the past two years
* General weakness/malaise (difficulty in walking, lack of autonomy, etc.). that substantially hinders participation in the study, regardless of their willingness to participate.
* Mental incapacity according to the investigator judgment.
* Not resident in the province in which the hospital is located.
* Not fluent in Spanish
* Allergy to iodinated contrast
* Morbid obesity (BMI> 40)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted in any of the participating ECOS hospitals with a diagnosis of COPD exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to new COPD exacerbation | One year
  From discharge of the current hospitalization, the time to a new COPD exacerbation will be estimated. The final aim of this study, descriptive, exploratory and hypothesis-generating, is to obtain a better understanding of the pathobiology of COPD exacerbations to eventually identify clinical correlations (biomarkers) that can help identify and diagnose them more accurately, and guide clinical practice for a more efficient way.

SECONDARY OUTCOMES:
Characterization and severity of pulmonary and systemic inflammation | One year
  Describe the biological characterization and severity of pulmonary and systemic inflammation, by means of presence/absence of inflamatory markers, their combination and their concentrations
Paired, Individual changes in pulmonary and systemic inflammation | One year
  Within individuals, characterization and severity of pulmonary and systemic inflammation, by means of presence/absence of inflamatory markers, their combination and their concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Noell G, Cosio BG, Faner R, Monso E, Peces-Barba G, de Diego A, Esteban C, Gea J, Rodriguez-Roisin R, Garcia-Nunez M, Pozo-Rodriguez F, Kalko SG, Agusti A. Multi-level differential network analysis of COPD exacerbations. Eur Respir J. 2017 Sep 27;50(3):1700075. doi: 10.1183/13993003.00075-2017. Print 2017 Sep. PMID 28954781